CLINICAL TRIAL: NCT01212952
Title: MC1082: A Phase I/II Trial of Pomalidomide (CC-4047), Bortezomib, and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Pomalidomide, Bortezomib, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1082; NCI-2010-01967 (Registry Identifier: NCI's CTRO); 10-001545 (Other: Mayo Clinic IRB); PO-MM-PI-0019 (Other: Celgene Protocol); MC1082 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2019-02

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Bortezomib; Dexamethasone; Calcium Dobesilate; Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral pomalidomide on days 1-21; bortezomib IV on days 1, 8, 15, 22; and oral dexamethasone on days 1, 8, 15, 22. Treatment repeats every 28 days for 8 courses. Patients then receive maintenance therapy comprising oral pomalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pomalidomide; Drug: bortezomib; Drug: dexamethasone; Other: laboratory biomarker analysis; Other: gene expression analysis

INTERVENTIONS:
Drug: pomalidomide — Given orally
  Other Names: CC-4047
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; Decaspray; DM; DXM
Other: laboratory biomarker analysis — Optional correlative studies
Other: gene expression analysis — Optional correlative studies

SUMMARY:
RATIONALE: Pomalidomide and bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bortezomib may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pomalidomide and bortezomib together with dexamethasone may kill more tumor cells. PURPOSE: This phase I/II trial is studying the side effects and best dose of bortezomib when given together with pomalidomide and dexamethasone and to see how well it works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of bortezomib in combination with pomalidomide and dexamethasone.

II. To evaluate the hematologic response rate (PR, VGPR, or CR) of pomalidomide, bortezomib and dexamethasone in patients with relapsed or refractory myeloma.

SECONDARY OBJECTIVES:

I. Time to progression.

II. To assess the toxicity of pomalidomide, bortezomib and dexamethasone in this patient population.

OUTLINE : This is a phase I, dose-escalation study of bortezomib followed by a phase II study. Patients receive oral pomalidomide on days 1-21; bortezomib IV on days 1, 8,15, 22; and oral dexamethasone on days 1, 8, 15, 22 . Treatment repeats every 28 days for 8 courses. Patients then receive maintenance therapy comprising oral pomalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Serum Creatinine =< 3 mg/dL
* Absolute neutrophil count >= 1000/uL
* Platelet count >= 75,000/uL
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * serum monoclonal protein >= 1.0 g/dL
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * monoclonal bone marrow plasmacytosis >= 30% (evaluable disease)
  * measurable plasmacytoma that has not been radiated
* ECOG Performance status (PS) 0, 1, or 2
* Previously treated relapsed or refractory multiple myeloma
* Patients must have received at least one prior therapy but no more than 4 therapies.

  * one or more of the prior regimens must have included lenalidomide and it has been determined the patient is refractory, resistant, or relapsed this therapy
  * prior bortezomib not required but if prior exposure, patients should not be refractory (Refractory means progression on therapy or within 60 days from the last dose of bortezomib.)
* Provide informed written consent
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide; FCBP must also agree to ongoing pregnancy testing
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy
* All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Willing and able to take aspirin or alternate prophylactic anticoagulation
* All previous cancer therapy, including chemotherapy, high dose corticosteroids, immune modulatory drugs or proteosome inhibitors must have been discontinued >= 2 weeks prior to study registration
* Any prior treatment with investigational agents must be discontinued >= 28 days prior to study registration
* Willing to abstain from donating blood during study participation and for 28 days after discontinuation of study drug
* Men must agree to abstain from donating semen or sperm during study participation and for 28 days after discontinuation of study drug
* Willingness to return to enrolling institution for follow-up

Exclusion Criteria:

* Concomitant high dose corticosteroids (concurrent use of corticosteroids); EXCEPTION: Patients may be on chronic steroids (maximum dose 20 mg/day prednisone equivalent) if they are being given for disorders other than myeloma, i.e., adrenal insufficiency, rheumatoid arthritis, etc
* Another malignancy undergoing active treatment with the exception of non melanoma skin cancer or in situ cervical or breast cancer
* Pregnant women or women of reproductive ability who are unwilling to use effective contraception
* Nursing women
* Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational: NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Active DVT or PE that has not been therapeutically anticoagulated
* Known positive for HIV or active hepatitis infection
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Known hypersensitivity to thalidomide or lenalidomide including development of erythema nodosum if characterized by a desquamating rash
* > grade 2 peripheral neuropathy
* Any prior use of pomalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Lacy, M.D., Study Chair — Mayo Clinic; Joseph R. Mikhael, M.D., Principal Investigator — Mayo Clinic; Vivek Roy, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Paludo J, Mikhael JR, LaPlant BR, Halvorson AE, Kumar S, Gertz MA, Hayman SR, Buadi FK, Dispenzieri A, Lust JA, Kapoor P, Leung N, Russell SJ, Dingli D, Go RS, Lin Y, Gonsalves WI, Fonseca R, Bergsagel PL, Roy V, Sher T, Chanan-Khan AA, Ailawadhi S, Stewart AK, Reeder CB, Richardson PG, Rajkumar SV, Lacy MQ. Pomalidomide, bortezomib, and dexamethasone for patients with relapsed lenalidomide-refractory multiple myeloma. Blood. 2017 Sep 7;130(10):1198-1204. doi: 10.1182/blood-2017-05-782961. Epub 2017 Jul 6. PMID 28684537

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1: Patients receive oral pomalidomide on days 1-21; bortezomib IV on days 1, 8, 15, 22; and oral dexamethasone on days 1, 8, 15, 22. Treatment repeats every 28 days for 8 courses. Patients then receive maintenance therapy comprising oral pomalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. 1.0 mg/m2 Bortezomib, 4 mg Pomalidomide, 40 mg Dexamethasone
- Phase 1 Dose Level 2; Phase 2 Dose Level 2: Patients receive oral pomalidomide on days 1-21; bortezomib IV on days 1, 8, 15, 22; and oral dexamethasone on days 1, 8, 15, 22. Treatment repeats every 28 days for 8 courses. Patients then receive maintenance therapy comprising oral pomalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. 1.3 mg/m2 Bortezomib, 4 mg Pomalidomide, 40 mg Dexamethasone
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 2 Dose Level 2
Started | 3 | 6 | 41
Completed | 3 | 6 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1; Dose Level 1; Phase 1; Dose Level 2; Phase 2; Dose Level 2: Patients receive oral pomalidomide on days 1-21; bortezomib IV on days 1, 8, 15, 22; and oral dexamethasone on days 1, 8, 15, 22. Treatment repeats every 28 days for 8 courses. Patients then receive maintenance therapy comprising oral pomalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1; Dose Level 1 | Phase 1; Dose Level 2 | Phase 2; Dose Level 2 | Total
Number analyzed (Participants) | 3 | 6 | 41 | 50
Age, Continuous [Median (Full Range); unit: years] | 63 [58 to 69] | 61 [45 to 73] | 66 [47 to 83] | 65.5 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 20 | 24
  Male | 3 | 2 | 21 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 3 | 5 | 39 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Find Maximum Tolerated Dose (MTD) of Bortezomib in Combination With Pomalidomide and Dexamethasone Out to 2.5 Years, by Count of Patients With Dose Limiting Toxicities.
Description: MTD is defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients).
Time Frame: 2.5 years
Population: The first 9 patients accrued(All Phase 1 patients) were evaluated for the MTD.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2
Number analyzed (Participants) | 3 | 6
Participants | 0 | 1
Statistical Analysis 1: Comparison: Phase 1 Dose Level 1 vs Phase 1 Dose Level 2; Test type: Other; Maximum Tolerated Dose (MTD) (mg/m^2) = 1.3 — Maximum Tolerated Dose Level is Dose Level 2 (1.3 mg/m^2 Bortezomib)

2. Primary Outcome: Number of Participants With a Hematologic Response (PR, VGPR, or CR)
Description: The number of participants who achieve PR, VGPR, or CR as defined by The International Myeloma Working Group uniform response criteria(2011). sCR: CR as defined below plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence. CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or > 90% reduction in serum M-protein plus urine M-protein level < 100 mg/24 h. PR: > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h. MR: NA. SD: Not meeting criteria for CR, VGPR, PR, or progressive disease. PD: Increase of > 25% from lowest response value in any one or more of the following: Serum M-component and/or (the absolute increase must be > 0.5 g/dL), Urine M-component and/or (the absolute increase must be > 200 mg/24 h)
Time Frame: 2.5 years
Measure: Count of Participants; unit: Participants
Groups:
- Phase I - Dose Level 1: Patients receive oral pomalidomide on days 1-21; bortezomib IV on days 1, 8, 15, 22; and oral dexamethasone on days 1, 8, 15, 22. Treatment repeats every 28 days for 8 courses. Patients then receive maintenance therapy comprising oral pomalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. 1.0 mg/m2 Bortezomib, 4 mg Pomalidomide, 40 mg Dexamethasone
- Phase I - Dose Level 2; Phase II: Patients receive oral pomalidomide on days 1-21; bortezomib IV on days 1, 8, 15, 22; and oral dexamethasone on days 1, 8, 15, 22. Treatment repeats every 28 days for 8 courses. Patients then receive maintenance therapy comprising oral pomalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. 1.3 mg/m2 Bortezomib, 4 mg Pomalidomide, 40 mg Dexamethasone
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase II
Number analyzed (Participants) | 3 | 6 | 41
Participants
  CR | 0 | 1 | 4
  PR | 0 | 1 | 17
  VGPR | 0 | 2 | 12
  SD | 1 | 0 | 5
  MR | 0 | 0 | 1
  sCR | 2 | 2 | 2

3. Secondary Outcome: Progression Free Survival
Description: The progression-free survival (PFS) time is defined as the time from registration to progression or death due to any cause. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. PD: Increase of > 25% from lowest response value in any one or more of the following: Serum M-component and/or (the absolute increase must be > 0.5 g/dL), Urine M-component and/or (the absolute increase must be > 200 mg/24 h)
Time Frame: 2.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase II
Number analyzed (Participants) | 3 | 6 | 41
months | 13.9 [2.8 to 22.9] | 18.1 [9.5 to NA] — The 95% confidence interval upper limit was not reached (i.e. insufficient number of events). | 10.7 [9.0 to 16.3]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Reported in Adverse Events section of the results
Time Frame: 2.5 years
Population: All participants combined in this analysis due to small numbers in Phase I portion.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase II
Number analyzed (Participants) | 3 | 6 | 41
Participants | 3 | 6 | 41

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Phase 1; Dose Level 1 | Phase 1; Dose Level 2 | Phase 2; Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 1/41
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/6 | 21/41
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1; Dose Level 1 (N=3) | Phase 1; Dose Level 2 (N=6) | Phase 2; Dose Level 2 (N=41)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 8 (11)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1; Dose Level 1 (N=3) | Phase 1; Dose Level 2 (N=6) | Phase 2; Dose Level 2 (N=41)
Anemia (Blood and lymphatic system disorders) | 3 (39) | 5 (55) | 39 (363)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (10) | 4 (19) | 29 (118)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (10) | 20 (100)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (20)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 3 (4)
Fatigue (General disorders) | 3 (29) | 6 (115) | 39 (436)
Fever (General disorders) | 0 (0) | 0 (0) | 3 (3)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 5 (11)
Lung infection (Infections and infestations) | 1 (1) | 2 (3) | 12 (20)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Creatinine increased (Investigations) | 1 (6) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (4) | 3 (9) | 16 (83)
Neutrophil count decreased (Investigations) | 3 (33) | 6 (81) | 41 (310)
Platelet count decreased (Investigations) | 2 (37) | 5 (41) | 36 (236)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 3 (33) | 6 (61) | 39 (291)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (7)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (37) | 6 (46) | 35 (346)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (3) | 1 (2) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT01212952/Prot_SAP_ICF_000.pdf